CLINICAL TRIAL: NCT06543290
Title: Azithromycin to Prevent Chorioamnionitis in Women Undergoing Induction of Labor, a Randomized Control Trial
Brief Title: Azithromycin Before Induction
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-33
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Infections
MeSH Terms: conditions — Infections | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: The investigators propose a double blinded randomized control trial of patients scheduled to undergo induction of labor at our institution. Enrolled patients will be randomized to receive a single dose of 2 grams Azithromycin or placebo. Induction will proceed per hospital protocols and the primary and secondary outcomes will be obtained from chart review after delivery and will end 6 weeks postpartum
Who Masked: Participant, Investigator
Masking Description: Pharmacy will have data set with participants idea and placebo vs study drug. All others will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin Arm (Active Comparator): Administration of 2 grams oral azithromycin (4 tablets of 500 mg) prior to the start of induction , once.
  Interventions: Drug: Azithromycin Pill
- Placebo Arm (Placebo Comparator): Administration of 4 magnesium oxide tablets prior to the start of induction , once.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin Pill — Azithromycin 2 grams to be administered prior to start of induction for those randomized to intervention group
  Arms: Azithromycin Arm
Drug: Placebo — 4 magnesium oxide tablets prior to the start of induction for those randomized to placebo
  Arms: Placebo Arm

SUMMARY:
This is a double blinded randomized control trial involving administration of 2 grams prophylactic azithromycin in third trimester patients undergoing induction of labor at our institution to demonstrate reduction in maternal and neonatal infection.

DETAILED DESCRIPTION:
Induction rates have more than tripled in the last quarter century, and even more in the past five years in light of evidence that the 39th week is the optimal gestational age for birth. Inductions are one of the most commonly performed medical procedures, and may span several days. One of the complications associated with induction include maternal infection, which includes chorioamnionitis, endometritis, pyelonephritis, neonatal infection, perineal and cesarean wound infections. There are many well-known risk factors for these infections that include longer duration of rupture of membrane, prolonged labor, nulliparity, internal monitoring, multiple vaginal examinations and several others. Well-established guidelines are available for treating infection once diagnosed, however the role of antibiotic prophylaxis to prevent infection in patients undergoing induction of labor is less clear. In this study, the investigators propose that administration of 2 grams oral azithromycin prior to the start of induction of labor will decrease rates of intrapartum and postpartum infections. Azithromycin is the ideal antibiotic to study in this trial since it is long acting, inexpensive, well tolerated, and has proven benefits in prior studies for prevention of obstetrical infection in cesarean deliveries and spontaneous labor. This is a double blinded randomized control trial involving administration of 2 grams prophylactic azithromycin in third trimester patients undergoing induction of labor at our institution to demonstrate reduction in maternal and neonatal infection. Decreasing rates of infection will improve both maternal and neonatal outcomes as well as decrease hospital length of stay and associated costs.

ELIGIBILITY:
Inclusion Criteria:

* • Third trimester of pregnancy defined as 28 0/7 weeks or more

  * Singleton pregnancy
  * Age 18-45
  * Induction of labor initiated for medical or obstetrical reason or electively over 39 weeks of gestation
  * No contraindication to vaginal delivery
  * Reassuring fetal heart rate tracing
  * Able and willing to provide informed consent

Exclusion Criteria:

* • Does not read or write in English or Spanish

  * Unable or unwilling to give informed consent
  * Use of antibiotic or antiviral agent within the last 7 days
  * Evidence of active infection at the time of initiation of induction (patients with rectovaginal group B streptococcus positive results will be allowed to participate as it is a colonizing organism, unless they show evidence of active infection)
  * Incarcerated Women
  * Active substance abuse
  * Age < 18

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Infection | Delivery and 6 weeks postpartum
  single oral dose of Azithromycin given prior to the start of induction of labor will decrease rates of composite infection

SECONDARY OUTCOMES:
Change in Infection | Delivery and 6 weeks postpartum
  single oral dose of azithromycin will also decrease rates of chorioamnionitis, endometritis, wound infection (both perineal and cesarean), neonatal infection and readmission rates, pyelonephritis, endomyometritis

CONTACTS AND LOCATIONS:
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Natality public-use data 2016-2018, on CDC WONDER Online Database. Division of Vital Statistics, 2020.
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Grobman WA, Caughey AB. Elective induction of labor at 39 weeks compared with expectant management: a meta-analysis of cohort studies. Am J Obstet Gynecol. 2019 Oct;221(4):304-310. doi: 10.1016/j.ajog.2019.02.046. Epub 2019 Feb 25. PMID 30817905
- [Background] Woodd SL, Montoya A, Barreix M, Pi L, Calvert C, Rehman AM, Chou D, Campbell OMR. Incidence of maternal peripartum infection: A systematic review and meta-analysis. PLoS Med. 2019 Dec 10;16(12):e1002984. doi: 10.1371/journal.pmed.1002984. eCollection 2019 Dec. PMID 31821329
- [Background] Tita AT, Andrews WW. Diagnosis and management of clinical chorioamnionitis. Clin Perinatol. 2010 Jun;37(2):339-54. doi: 10.1016/j.clp.2010.02.003. PMID 20569811
- [Background] Pierce SL, Peck JD, Zornes C, Standerfer E, Edwards RK. Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term: a pilot randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Sep;4(5):100681. doi: 10.1016/j.ajogmf.2022.100681. Epub 2022 Jun 18. PMID 35728781
- [Background] Tita AT, Szychowski JM, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Abramovici A, Ambalavanan N, Cutter G, Andrews W; C/SOAP Trial Consortium. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2016 Sep 29;375(13):1231-41. doi: 10.1056/NEJMoa1602044. PMID 27682034